CLINICAL TRIAL: NCT06323304
Title: Evaluating Efficacy and Safety of Auricular Acupressure in Treating Allergic Rhinitis: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Auricular Acupressure in Treating Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 701/HDDD-DHYD
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Itching; Runny Nose; Sneezing; Nasal Congestion
Keywords: Allergic rhinitis; Auricular acupressure therapy; Traditional medicine
MeSH Terms: conditions — Pruritus; Rhinorrhea; Sneezing; Nasal Obstruction; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind method (Participant, Investigator, Outcome assessor) Participants will be blinded to their randomization assignment, either to the intervention group or the control group. Sham acupressure therapy will be performed at acupoints that have no therapeutic effect on allergic rhinitis, and the procedures will be similar to auricular pressure therapy. Both groups will be treated with fluticasone propionate nasal spray, which is the standard treatment.
  The physician who perform auricular acupressure therapy or sham acupressure therapy will be aware of the intervention assignment for each group, but they will not be involved in data analysis or outcome assessment. The data analysts and outcome assessors will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupressure + fluticasone propionate nasal spray (Experimental): Auricular acupressure therapy (AAT) once a week on the left ear for a total of four weeks (4 sessions). Fluticasone propionate nasal spray will be used whenever symptoms occur.
  Interventions: Other: Auricular acupressure; Other: Standard treatment
- Sham acupressure + fluticasone propionate nasal spray (Sham Comparator): Sham acupressure therapy (SAT) once a week on the left ear for a total of four weeks (4 sessions). Fluticasone propionate nasal spray will be used whenever symptoms occur.
  Interventions: Other: Sham acupressure; Other: Standard treatment

INTERVENTIONS:
Other: Auricular acupressure — Auricular acupressure therapy will be performed once a week for 4 weeks using Vaccaria seeds, which is an herb in traditional medicine. The acupoints on the ear that will be treated with auricular acupressure therapy are Shenmen (TF4), Internal nose (TG4), Lung (CO14), Wind stream (SF1,2i), Adrenal gland (TG2p). These acupoints are believed to be effective in the treatment of allergic rhinitis. The patches will be kept on the auricle for one week.
  Arms: Auricular acupressure + fluticasone propionate nasal spray
Other: Sham acupressure — Sham acupressure therapy will be performed once a week for 4 weeks using Vaccaria seeds. The acupoints that will be treated with auricular acupressure therapy are Helix 2 (HX10), Shoulder (SF4), Clavicle (SF6), Anus (HX5) and Tooth (LO1). These acupoints are not used to treat allergic immune-related problems or respiratory diseases. The patches will be kept on the auricle for one week.
  Arms: Sham acupressure + fluticasone propionate nasal spray
Other: Standard treatment — Standard treatment, continuously administered over the 4-week intervention period, involves standard doses of fluticasone propionate nasal spray as needed, and lifestyle modifications.

SUMMARY:
Allergic rhinitis (AR) is a global health problem affecting approximately 10% to 40% of the population worldwide, with an increasing trend. It significantly impacts health and quality of life. Current treatments for AR include allergen avoidance, symptom-relieving medications, anti-inflammatory therapy, and allergen-specific immunotherapy. However, many patients still experience uncontrolled symptoms despite these approaches, either as monotherapy or in combination, along with medication side effects such as drowsiness, dry eyes, nasal mucosal damage, and immunosuppression.

Auricular acupressure therapy (AAT) utilizes ear acupoints by applying pressure with ear seeds. The neurobiological mechanisms of AAT on the human body have gained increasing attention in clinical and experimental studies, involving anti-inflammatory, antioxidant, and immunomodulatory effects. Its efficacy has been recognized, becoming a potential alternative therapy for various conditions such as sleep disorders, obesity, and chronic pain. Previous clinical studies have reported the efficacy and safety of AAT in treating AR. However, the primary outcomes of these studies remain inconsistent and lack specific criteria for evaluating AR treatment efficacy.

This study aims to investigate the efficacy and safety of AAT in treating AR based on the ARIA guideline 2019 treatment efficacy criteria. It will provide a basis for applying AAT as a complementary approach in the multimodal treatment of AR.

DETAILED DESCRIPTION:
Patients with allergic rhinitis who have typical symptoms such as nasal itching, runny nose, sneezing, nasal congestion, and are indicated for corticosteroid nasal spray according to the ARIA 2019 diagnostic and treatment guidelines will be registered for this study. They will then be randomly assigned to two groups: Intervention group (auricular acupressure therapy + fluticasone propionate nasal spray), and control group (sham auricular acupressure therapy + fluticasone propionate nasal spray). The allocation ratio for the two groups is 1:1.

The intervention period for both groups is four weeks. Auricular acupressure therapy or sham acupressure therapy will be performed every week. Fluticasone propionate nasal spray will be used whenever symptoms occur. Patients will also be encouraged to adjust their lifestyle and living environment.

Data on the severity of allergic rhinitis symptoms (including nasal itching, sneezing, runny nose, nasal congestion, eye symptoms, and headache), the Rhinitis Quality of Life Questionnaire (RQLQ), and side effects of auricular acupressure therapy will be recorded before the study and weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with allergic rhinitis according to the ARIA 2019 (Allergic Rhinitis and its Impact on Asthma) diagnostic criteria, must be between 18 and 60 years old.
* Must have had typical symptoms of allergic rhinitis for at least 2 years.
* Must provide written informed consent to participate in the study.
* Must be mentally alert and able to communicate effectively.
* Must have vital signs within normal limits (pulse, blood pressure, temperature, respiratory rate, SpO2).
* Must not have any other chronic diseases, including respiratory diseases (asthma, pneumonia, chronic obstructive pulmonary disease, etc.), thyroid disease, autonomic nervous system disorders, hypertension, or diabetes, as determined by medical history.
* Must not have any knowledge of auricular therapy.

Exclusion Criteria:

* Have used decongestants, antihistamines, anticholinergics, or oral corticosteroids within the past 1 week.
* Have undergone auricular acupuncture, auricular acupressure, or other forms of acupuncture for the treatment of other respiratory diseases within the past 6 months.
* Have used stimulants (alcohol, beer, coffee, tobacco) within 24 hours of the study.
* Lesions (scars, tears, scratches, bites) on the left auricle.
* Allergic rhinitis with secondary infection, acute sinusitis or acute exacerbation of chronic sinusitis, or chronic sinusitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The change of nasal and non nasal symptom scores | Assessments were conducted before intervention and after each intervention week throughout the four weeks (Week 0, Week 1, Week 2, Week 3, Week 4)
  Symptom scores will be assessed based on a visual analogue scale (VAS). It usually consists of a 100 mm line anchored at each end by descriptors.

SECONDARY OUTCOMES:
The change of Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) score | Assessments were conducted before intervention and after each intervention week throughout the four weeks (Week 0, Week 1, Week 2, Week 3, Week 4)
  The RQLQ consists of 28 items. Participants will be requested to express their agreement using a Likert-type scale that ranges from 0=not troubled to 6=extremely troubled. The RQLQ score is calculated by taking the sum of the scores for all question. The higher the score, the more impaired the quality of life.
The change of relief medication usage | Assessments were conducted after each intervention week throughout the four weeks (Week 1, Week 2, Week 3, Week 4)
  The number of times fluticasone propionate nasal spray is used is recorded each week by asking the patient.
Proportion of intervention-related adverse events | Up to four weeks
  While auricular acupressure is generally considered safe, some patients may experience minor side effects at the application site. These can include temporary pain, discomfort, itching, redness, or minor inflammation. Rarely, more serious complications like chondritis, dizziness, nausea, or allergic reactions may occur. The study will closely monitor and document any unexpected adverse events associated with the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Bousquet JJ, Schunemann HJ, Togias A, Erhola M, Hellings PW, Zuberbier T, Agache I, Ansotegui IJ, Anto JM, Bachert C, Becker S, Bedolla-Barajas M, Bewick M, Bosnic-Anticevich S, Bosse I, Boulet LP, Bourrez JM, Brusselle G, Chavannes N, Costa E, Cruz AA, Czarlewski W, Fokkens WJ, Fonseca JA, Gaga M, Haahtela T, Illario M, Klimek L, Kuna P, Kvedariene V, Le LTT, Larenas-Linnemann D, Laune D, Lourenco OM, Menditto E, Mullol J, Okamoto Y, Papadopoulos N, Pham-Thi N, Picard R, Pinnock H, Roche N, Roller-Wirnsberger RE, Rolland C, Samolinski B, Sheikh A, Toppila-Salmi S, Tsiligianni I, Valiulis A, Valovirta E, Vasankari T, Ventura MT, Walker S, Williams S, Akdis CA, Annesi-Maesano I, Arnavielhe S, Basagana X, Bateman E, Bedbrook A, Bennoor KS, Benveniste S, Bergmann KC, Bialek S, Billo N, Bindslev-Jensen C, Bjermer L, Blain H, Bonini M, Bonniaud P, Bouchard J, Briedis V, Brightling CE, Brozek J, Buhl R, Buonaiuto R, Canonica GW, Cardona V, Carriazo AM, Carr W, Cartier C, Casale T, Cecchi L, Cepeda Sarabia AM, Chkhartishvili E, Chu DK, Cingi C, Colgan E, de Sousa JC, Courbis AL, Custovic A, Cvetkosvki B, D'Amato G, da Silva J, Dantas C, Dokic D, Dauvilliers Y, Dedeu A, De Feo G, Devillier P, Di Capua S, Dykewickz M, Dubakiene R, Ebisawa M, El-Gamal Y, Eller E, Emuzyte R, Farrell J, Fink-Wagner A, Fiocchi A, Fontaine JF, Gemicioglu B, Schmid-Grendelmeir P, Gamkrelidze A, Garcia-Aymerich J, Gomez M, Gonzalez Diaz S, Gotua M, Guldemond NA, Guzman MA, Hajjam J, O'B Hourihane J, Humbert M, Iaccarino G, Ierodiakonou D, Illario M, Ivancevich JC, Joos G, Jung KS, Jutel M, Kaidashev I, Kalayci O, Kardas P, Keil T, Khaitov M, Khaltaev N, Kleine-Tebbe J, Kowalski ML, Kritikos V, Kull I, Leonardini L, Lieberman P, Lipworth B, Lodrup Carlsen KC, Loureiro CC, Louis R, Mair A, Marien G, Mahboub B, Malva J, Manning P, De Manuel Keenoy E, Marshall GD, Masjedi MR, Maspero JF, Mathieu-Dupas E, Matricardi PM, Melen E, Melo-Gomes E, Meltzer EO, Menditto E, Mercier J, Miculinic N, Mihaltan F, Milenkovic B, Moda G, Mogica-Martinez MD, Mohammad Y, Montefort S, Monti R, Morais-Almeida M, Mosges R, Munter L, Muraro A, Murray R, Naclerio R, Napoli L, Namazova-Baranova L, Neffen H, Nekam K, Neou A, Novellino E, Nyembue D, O'Hehir R, Ohta K, Okubo K, Onorato G, Ouedraogo S, Pali-Scholl I, Palkonen S, Panzner P, Park HS, Pepin JL, Pereira AM, Pfaar O, Paulino E, Phillips J, Picard R, Plavec D, Popov TA, Portejoie F, Price D, Prokopakis EP, Pugin B, Raciborski F, Rajabian-Soderlund R, Reitsma S, Rodo X, Romano A, Rosario N, Rottem M, Ryan D, Salimaki J, Sanchez-Borges MM, Sisul JC, Sole D, Somekh D, Sooronbaev T, Sova M, Spranger O, Stellato C, Stelmach R, Suppli Ulrik C, Thibaudon M, To T, Todo-Bom A, Tomazic PV, Valero AA, Valenta R, Valentin-Rostan M, van der Kleij R, Vandenplas O, Vezzani G, Viart F, Viegi G, Wallace D, Wagenmann M, Wang Y, Waserman S, Wickman M, Williams DM, Wong G, Wroczynski P, Yiallouros PK, Yorgancioglu A, Yusuf OM, Zar HJ, Zeng S, Zernotti M, Zhang L, Zhong NS, Zidarn M; ARIA Study Group; MASK Study Group. Next-generation ARIA care pathways for rhinitis and asthma: a model for multimorbid chronic diseases. Clin Transl Allergy. 2019 Sep 9;9:44. doi: 10.1186/s13601-019-0279-2. eCollection 2019. PMID 31516692
- [Background] Dykewicz MS, Wallace DV, Amrol DJ, Baroody FM, Bernstein JA, Craig TJ, Dinakar C, Ellis AK, Finegold I, Golden DBK, Greenhawt MJ, Hagan JB, Horner CC, Khan DA, Lang DM, Larenas-Linnemann DES, Lieberman JA, Meltzer EO, Oppenheimer JJ, Rank MA, Shaker MS, Shaw JL, Steven GC, Stukus DR, Wang J; Chief Editor(s):; Dykewicz MS, Wallace DV; Joint Task Force on Practice Parameters:; Dinakar C, Ellis AK, Golden DBK, Greenhawt MJ, Horner CC, Khan DA, Lang DM, Lieberman JA, Oppenheimer JJ, Rank MA, Shaker MS, Stukus DR, Wang J; Workgroup Contributors:; Dykewicz MS, Wallace DV, Amrol DJ, Baroody FM, Bernstein JA, Craig TJ, Finegold I, Hagan JB, Larenas-Linnemann DES, Meltzer EO, Shaw JL, Steven GC. Rhinitis 2020: A practice parameter update. J Allergy Clin Immunol. 2020 Oct;146(4):721-767. doi: 10.1016/j.jaci.2020.07.007. Epub 2020 Jul 22. PMID 32707227
- [Background] Nogier R. History of Auriculotherapy: Additional Information and New Developments. Med Acupunct. 2021 Dec 1;33(6):410-419. doi: 10.1089/acu.2021.0075. Epub 2021 Dec 16. PMID 34976274
- [Background] Rao YQ, Han NY. [Therapeutic effect of acupuncture on allergic rhinitis and its effects on immunologic function]. Zhongguo Zhen Jiu. 2006 Aug;26(8):557-60. Chinese. PMID 16941973
- [Background] Zhong J, Liu S, Lai D, Lu T, Shen Y, Gong Q, Li P, Zhang Q. Ear Acupressure for Allergic Rhinitis: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2021 May 3;2021:6699749. doi: 10.1155/2021/6699749. eCollection 2021. PMID 34007299
- [Background] Zhang CS, Xia J, Zhang AL, Yang AW, Thien F, Li Y, Wu D, Cai J, DaCosta C, Xue CC. Ear acupressure for perennial allergic rhinitis: A multicenter randomized controlled trial. Am J Rhinol Allergy. 2014 Jul-Aug;28(4):e152-7. doi: 10.2500/ajra.2014.28.4081. PMID 25197908
- [Background] Butt MF, Albusoda A, Farmer AD, Aziz Q. The anatomical basis for transcutaneous auricular vagus nerve stimulation. J Anat. 2020 Apr;236(4):588-611. doi: 10.1111/joa.13122. Epub 2019 Nov 19. PMID 31742681
- [Background] Hou PW, Hsu HC, Lin YW, Tang NY, Cheng CY, Hsieh CL. The History, Mechanism, and Clinical Application of Auricular Therapy in Traditional Chinese Medicine. Evid Based Complement Alternat Med. 2015;2015:495684. doi: 10.1155/2015/495684. Epub 2015 Dec 28. PMID 26823672
- [Background] Feng L, Lin L, Wang S, Zhao X, Dai Q, Wang L, Yang Y, Xu L, Liu Y, An L, Shen C. Clinical practice guidelines for the treatment of allergic rhinitis in children with traditional Chinese medicine. Anat Rec (Hoboken). 2021 Nov;304(11):2592-2604. doi: 10.1002/ar.24718. Epub 2021 Jul 29. PMID 34323398
- [Background] Tan JY, Molassiotis A, Wang T, Suen LK. Adverse events of auricular therapy: a systematic review. Evid Based Complement Alternat Med. 2014;2014:506758. doi: 10.1155/2014/506758. Epub 2014 Nov 10. PMID 25435890
- [Derived] Le NC, Bui MP, Trinh DT. Evaluating efficacy and safety of auricular acupressure in treating allergic rhinitis: A randomized controlled trial. Integr Med Res. 2025 Sep;14(3):101177. doi: 10.1016/j.imr.2025.101177. Epub 2025 Jun 9. PMID 40677297
- See also: Related Info — https://www.who.int/publications/i/item/9789240042322